CLINICAL TRIAL: NCT04705402
Title: A Prospective, Randomized, Double Blinded, Placebo Control Trial to Evaluate Efficacy of Intravenous Mannitol Use During Cadaveric Kidney Transplantation Prior to Kidney Reperfusion
Brief Title: Mannitol Use During Cadaveric Kidney Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0826-20-RMC
Record Dates: First submitted 2021-01-10; First posted 2021-01-12 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Renal Dialysis
MeSH Terms: interventions — Mannitol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients randomized to receive the treatment arm of mannitol. (Experimental): The mannitol solution used in the hospital contain 18% mannitol in 500ml solution. An equivocal volume of 2.8 cc / kg body weight, which will be given intravenously with the use of an Ivac pump, infused for a duration of 15 minutes through an existing peripheral intravenous access catheter within 15-30 minutes prior to renal artery reperfusion
  Interventions: Drug: Mannitol
- (Control arm) Study participants will receive a 0.9% saline solution (Placebo Comparator): (Control arm) Study participants randomized to this arm will receive a 0.9% saline solution at a dose of 2.8 cc / kg, infused within 15-30 minutes prior to renal artery reperfusion through an existing intravenous access catheter (either through an central or peripheral intravenous infusion).
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Mannitol — Mannitol (Israeli Brand Name: Osmitrol) is in the osmotic diuretic pharmacologic categoryaccording to the American Hospital Formulary Service (AHFS) database. . During the procedure, volume of 2.8 cc / kg body weight of the solution bag (either mannitol or saline 0.9%) will be given. The bag itself will be covered so it cannot be identified which solution is in it and marked per patient.
  Mannitol is injected by intravenous infusion using an I-vac pump and infused over 15 minutes.
  Arms: Patients randomized to receive the treatment arm of mannitol.
Drug: Saline — Study participants randomized to this arm will receive a 0.9% saline solution at a dose of 2.8 cc / kg, infused within 15-30 minutes prior to renal artery reperfusion through an existing intravenous access catheter (either through an central or peripheral intravenous infusion).
  Arms: (Control arm) Study participants will receive a 0.9% saline solution

SUMMARY:
We propose a placebo controlled randomized study on the use of mannitol as an agent to protect against delayed graft function, during the surgical procedure of kidney transplantation from a cadaver. Patients undergoing kidney transplantation for the treatment of end stage kidney disease will be randomized in a ratio of 1:1 to receive either intravenous mannitol or saline during their procedure, administered prior to renal artery clamp release and reperfusion of the kidney. Changes in renal function following surgery and the incidence and duration of delayed graft function (DGF) will be monitored using calculated glomerular filtration rate (eGFR) and the need for dialysis performed post-operatively, as part of routine standard of care. Additionally biological samples will be collected and analyzed for use of a non invasive biomarker for delayed graft function.

DETAILED DESCRIPTION:
This study is a prospective randomized double-blind placebo-controlled trial comparing renal function outcomes in patients undergoing cadaver donor renal transplant for end stage kidney failure. Patients will be randomized to receive 0.5 g / kg body weight, of mannitol or saline 0.9% as an intravenous infusion to be initiated and be completely infused within 15-30 minutes prior to vascular clamp removal of the transplanted renal artery.

Prior to surgery, all study participants will receive standard departmental treatment as all other patients undergoing a kidney transplantation from a cadaver.

Upon arrival to the operating room patients will be placed supine on the operating room table, and will be connected to an anesthesia monitor which will include monitoring the HR, blood pressure, saturation, temperature and ECG as standard departmental procedure. After connecting the participant to the anesthesia monitor an IV line will be inserted, as is standard clinical practice. In addition, venous central line catheter for central venous pressure monitoring and specific inotropic drugs infusion, as well as arterial line catheter for blood pressure monitoring, will be initialized upon anesthesiologist team decision The technique of kidney transplantation is well-standardized . None of the techniques utilized in the study are considered experimental and all are considered standard therapeutic options for a patient undergoing cadaveric donor kidney transplantation. The procedures are performed under general anesthesia with non-invasive intraoperative vital sign monitoring, as is standard departmental practice. Study participation will not affect anesthesia method or protocol treatment in anyway.

Upon study enrollment patients will be randomized in 1:1 ratio for study arm treatment/control. The perioperative team, investigator and patient will be blinded to the intervention.

Study arm: Patients randomized to receive the treatment arm will receive 0.5 g / kg body weight of mannitol. The mannitol solution used in the hospital contain 18% mannitol in 500ml solution. An equivocal volume of 2.8 cc / kg body weight, which will be given intravenously with the use of an Ivac pump, infused for a duration of 15 minutes through an existing peripheral intravenous access catheter within 15-30 minutes prior to renal artery reperfusion.

The placebo arm (Control arm) Study participants randomized to this arm will receive a 0.9% saline solution at a dose of 2.8 cc / kg, infused within 15-30 minutes prior to renal artery reperfusion through an existing intravenous access catheter (either through an central or peripheral intravenous infusion).

Following receiving the study drug, either mannitol or saline, patients will receive 80 mg furosemide, which will be given intravenously.

Fluid management throughout the kidney transplant surgery for all study participants will consist as follows:

* Upon arrival to the operating room, immediately following IV insertion, all patients will receive an IV infusion of Plasma-Lyte as it is a standard protocol at our institute for kidney transplant surgery.
* After induction of anesthesia, the patient will receive Plasma-Lyte solution at a rate of 8 cc / kg body weight per hour.
* At this stage of the procedure, before reperfusion of the transplanted kidney, the purpose of this fluid management is intended to maintain a minimum systolic blood pressure of 90-100mmHg.
* At 30 to 15 minutes before reperfusion, in purpose to let the transplanted kidney get better opening conditions, the target blood pressure is elevated to an mean arterial pressure (MAP) of not less than 100 mmHg. In order to achieve that, additional 1000 cc of Plasma-Lyte will be given to the patient 30 to 15 minutes before re-perfusion. In addition, small boluses (each 0.1 mg) of Phenylephrine will be given as needed to maintain that MAP.
* Thereafter, and until the end of the operation, the fluid management will be titrated according to the patient's blood pressure, ensuring that systolic blood pressure does not fall below 120 mmHG, as the common departmental protocol in such surgeries. In occasions of hypotension, a bolus of 250 cc Plasma-Lyte will be given to increase the blood pressure.
* If there is insufficient response to repeat boluses, vasopressors (phenylephrine, ephedrine or noradrenaline) will be given at the discretion of the anesthesiologist.
* Episodes of hypotension not responsive to intravenous fluids will be treated with intravenous vasopressors (phenylephrine, ephedrine or noradrenaline as needed) at the discretion of the anesthesiologist. The provision of these drugs will be documented individually in the study report for each patient, as is common clinical practice.
* After surgery, in the post anesthesia care unit (PACU), the patient will receive 80 cc / hour of Plasma-Lyte or 120% of urine output if urine output exceeds 80 cc. Patients are regularly supervised in PACU for 2-4 hours after the end of the operation and then transferred to the department of organ transplantation. In cases of need for dialysis or prolonged ventilation, they stay at PACU.
* The fluid management for the postoperative days are as standard regimen in our center which consists of giving the patient full fluid replacement at POD1 - including urine output and drains output. On the next post-operative days, we replace 80% of urine output in IV fluids and oral intake together.

Additionally blood and urine samples maybe collected from some of the patients (In the event that it is possible) at the following different timelines:

Immediately before administering mannitol Immediately after administering mannitol 24 hours after transplant 7 days after transplant, These biological samples will be collected and analyzed to asses the presence of proteins, exosomes , cytokines that can be used as a non invasive biomarker for delayed graft function.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients on the list of cadaveric donor kidney transplantation

Exclusion Criteria:

* Allergy to mannitol
* Allergy to furosemide
* Combined major surgical cases that may include transplantation of another organ on the same time, such as liver.
* Severe congestive heart failure (ejection fraction < 30%)
* Patients with coagulation disorders.
* Patients who are not able to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of dialysis after surgery | within 7 days postoperatively
Urine Output ml per day | Within 7 days postoperatively.
Creatinine value | All 7 days postoperatively

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lugo-Baruqui JA, Ayyathurai R, Sriram A, Pragatheeshwar KD. Use of Mannitol for Ischemia Reperfusion Injury in Kidney Transplant and Partial Nephrectomies-Review of Literature. Curr Urol Rep. 2019 Jan 26;20(1):6. doi: 10.1007/s11934-019-0868-6. PMID 30685826
- [Background] Gagandeep S, Matsuoka L, Mateo R, Cho YW, Genyk Y, Sher L, Cicciarelli J, Aswad S, Jabbour N, Selby R. Expanding the donor kidney pool: utility of renal allografts procured in a setting of uncontrolled cardiac death. Am J Transplant. 2006 Jul;6(7):1682-8. doi: 10.1111/j.1600-6143.2006.01386.x. PMID 16827871
- [Background] Foroutan F, Friesen EL, Clark KE, Motaghi S, Zyla R, Lee Y, Kamran R, Ali E, De Snoo M, Orchanian-Cheff A, Ribic C, Treleaven DJ, Guyatt G, Meade MO. Risk Factors for 1-Year Graft Loss After Kidney Transplantation: Systematic Review and Meta-Analysis. Clin J Am Soc Nephrol. 2019 Nov 7;14(11):1642-1650. doi: 10.2215/CJN.05560519. Epub 2019 Sep 20. PMID 31540931
- [Background] de Sandes-Freitas TV, Felipe CR, Aguiar WF, Cristelli MP, Tedesco-Silva H, Medina-Pestana JO. Prolonged Delayed Graft Function Is Associated with Inferior Patient and Kidney Allograft Survivals. PLoS One. 2015 Dec 17;10(12):e0144188. doi: 10.1371/journal.pone.0144188. eCollection 2015. PMID 26679933
- [Background] Dawidson IJ, Sandor ZF, Coorpender L, Palmer B, Peters P, Lu C, Sagalowsky A, Risser R, Willms C. Intraoperative albumin administration affects the outcome of cadaver renal transplantation. Transplantation. 1992 Apr;53(4):774-82. doi: 10.1097/00007890-199204000-00014. PMID 1566343
- [Background] Willms CD, Dawidson IJ, Dickerman R, Drake D, Sandor ZF, Trevino G. Intraoperative blood volume expansion induces primary function after renal transplantation: a study of 96 paired cadaver kidneys. Transplant Proc. 1991 Feb;23(1 Pt 2):1338-9. No abstract available. PMID 1989234
- [Background] Lewis SR, Pritchard MW, Evans DJ, Butler AR, Alderson P, Smith AF, Roberts I. Colloids versus crystalloids for fluid resuscitation in critically ill people. Cochrane Database Syst Rev. 2018 Aug 3;8(8):CD000567. doi: 10.1002/14651858.CD000567.pub7. PMID 30073665
- [Background] Weimar W, Geerlings W, Bijnen AB, Obertop H, van Urk H, Lameijer LD, Wolff ED, Jeekel J. A controlled study on the effect of mannitol on immediate renal function after cadaver donor kidney transplantation. Transplantation. 1983 Jan;35(1):99-101. No abstract available. PMID 6401883
- [Background] Tiggeler RG, Berden JH, Hoitsma AJ, Koene RA. Prevention of acute tubular necrosis in cadaveric kidney transplantation by the combined use of mannitol and moderate hydration. Ann Surg. 1985 Feb;201(2):246-51. doi: 10.1097/00000658-198502000-00020. PMID 3918517
- [Background] von Moos S, Akalin E, Mas V, Mueller TF. Assessment of Organ Quality in Kidney Transplantation by Molecular Analysis and Why It May Not Have Been Achieved, Yet. Front Immunol. 2020 May 12;11:833. doi: 10.3389/fimmu.2020.00833. eCollection 2020. PMID 32477343
- [Background] Reiterer C, Hu K, Sljivic S, Falkner von Sonnenburg M, Fleischmann E, Kainz A, Kabon B. Mannitol and renal graft injury in patients undergoing deceased donor renal transplantation - a randomized controlled clinical trial. BMC Nephrol. 2020 Jul 28;21(1):307. doi: 10.1186/s12882-020-01961-z. PMID 32723374
- [Background] Gremmels H, de Jong OG, Toorop RJ, Michielsen L, van Zuilen AD, Vlassov AV, Verhaar MC, van Balkom BWM. The Small RNA Repertoire of Small Extracellular Vesicles Isolated From Donor Kidney Preservation Fluid Provides a Source for Biomarker Discovery for Organ Quality and Posttransplantation Graft Function. Transplant Direct. 2019 Aug 12;5(9):e484. doi: 10.1097/TXD.0000000000000929. eCollection 2019 Sep. PMID 31579812
- [Background] Siew ED, Ware LB, Ikizler TA. Biological markers of acute kidney injury. J Am Soc Nephrol. 2011 May;22(5):810-20. doi: 10.1681/ASN.2010080796. Epub 2011 Apr 14. PMID 21493774
- [Background] Tataruch-Weinert D, Musante L, Kretz O, Holthofer H. Urinary extracellular vesicles for RNA extraction: optimization of a protocol devoid of prokaryote contamination. J Extracell Vesicles. 2016 Jun 24;5:30281. doi: 10.3402/jev.v5.30281. eCollection 2016. PMID 27345058
- [Background] Feng Y, Lv LL, Wu WJ, Li ZL, Chen J, Ni HF, Zhou LT, Tang TT, Wang FM, Wang B, Chen PS, Crowley SD, Liu BC. Urinary Exosomes and Exosomal CCL2 mRNA as Biomarkers of Active Histologic Injury in IgA Nephropathy. Am J Pathol. 2018 Nov;188(11):2542-2552. doi: 10.1016/j.ajpath.2018.07.017. Epub 2018 Aug 22. PMID 30142333